CLINICAL TRIAL: NCT00005900
Title: Study of Pulmonary Complications in Pediatric Patients With Storage Disorders Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fairview University Medical Center (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/15111; UMN-MT-1999-18; UMN-MT-9818
Record Dates: First submitted 2000-06-02; First posted 2000-06-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-10

CONDITIONS: I Cell Disease; Fucosidosis; Globoid Cell Leukodystrophy; Adrenoleukodystrophy; Mannosidosis; Niemann-Pick Disease; Pulmonary Complications; Mucopolysaccharidosis I; Mucopolysaccharidosis VI; Metachromatic Leukodystrophy; Gaucher's Disease; Wolman Disease
Keywords: Gaucher's disease; I cell disease; Niemann-Pick disease; Wolman disease; adrenoleukodystrophy; disease-related problem/condition; fucosidosis; genetic diseases and dysmorphic syndromes; globoid cell leukodystrophy; inborn errors of metabolism; mannosidosis; metachromatic leukodystrophy; mucopolysaccharidosis; mucopolysaccharidosis I; mucopolysaccharidosis VI; oncologic disorders; pulmonary complications; rare disease; sphingolipidoses
MeSH Terms: conditions — Mucolipidoses; Fucosidosis; Leukodystrophy, Globoid Cell; Adrenoleukodystrophy; Mannosidase Deficiency Diseases; Niemann-Pick Diseases; Mucopolysaccharidosis I; Mucopolysaccharidosis VI; Leukodystrophy, Metachromatic; Gaucher Disease; Wolman Disease; Genetic Diseases, Inborn; Metabolism, Inborn Errors; Mucopolysaccharidoses; Rare Diseases; Sphingolipidoses

SUMMARY:
OBJECTIVES: I. Evaluate bronchoalveolar lavage fluid and serum obtained from pediatric patients with storage disorders prior to allogeneic hematopoietic stem cell transplantation (HSCT) for the presence of proinflammatory cytokines and for the production of nitric oxide by alveolar macrophages to identify possible risk factors for pulmonary complications.

II. Investigate the underlying mechanism for the development of significant pulmonary complications in these patients during HSCT.

III. Evaluate bronchoalveolar lavage fluid and serum obtained from these same patients at the time a pulmonary complication develops post-HSCT, or at 60 days post-HSCT if there has been no pulmonary complications.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients undergo bronchoscopy with bronchoalveolar lavage (BAL) prior to allogeneic hematopoietic stem cell transplantation (HSCT). ELISA assays for cytokines are performed. Patients are followed post-HSCT for the development of transplant related pulmonary complications. A repeat bronchoscopy with BAL is performed at the time pulmonary complications develop or at day 60 post-HSCT if no complications develop. Cytokine assays are repeated.

ELIGIBILITY:
* Diagnosis of an inborn error of metabolism eligible for allogeneic hematopoietic stem cell transplantation on protocol UMN-MT-1995-01

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 1999-08

CONTACTS AND LOCATIONS:
Overall Officials: K. Scott Baker, Study Chair — Fairview University Medical Center
Locations (1):
- Fairview University Medical Center, Minneapolis, Minnesota, United States